CLINICAL TRIAL: NCT03446885
Title: Efficacy of Lisdexamfetamine Dimesylate for Promoting Occupational Success in Young Adults With Attention-deficit/Hyperactivity Disorder
Brief Title: Efficacy of Lisdexamfetamine Dimesylate for Promoting Occupational Success in Young Adults With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gregory Fabiano (Other)
Responsible Party: Sponsor-Investigator, Gregory Fabiano, Professor, State University of New York at Buffalo
Organization: State University of New York at Buffalo (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IIR-USA-001277
Record Dates: First submitted 2017-08-31; First posted 2018-02-27 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Intervention Model Description: All participants received placebo and 40 mg Vyvanse in a cross-over design. Order of administration was randomly assigned and counter-balanced across participants
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lab visit 1 (Experimental): 40 mg of Vyvanse administered q.a.m. or Placebo administered in random, counter-balanced fashion.
  Interventions: Drug: Lisdexamfetamine Dimesylate 40 MG; Drug: Placebo
- Lab visit 2 (Experimental): 40 mg of Vyvanse administered q.a.m. or Placebo administered in random, counter-balanced fashion.
  Interventions: Drug: Lisdexamfetamine Dimesylate 40 MG; Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate 40 MG — Lisdexamfetamine Dimesylate 40 MG administered orally
Drug: Placebo — Placebo capsule administered orally

SUMMARY:
There has been little research on the third area of impairment noted in the Diagnostic and Statistical Manual of Mental Disorders - "occupational functioning." Individuals with ADHD experience job-related impairments including a greater likelihood of being unemployed and not enrolled in school and for those that were employed they were in a lower status occupation, relative to typically-developing comparison peers. The current literature on analogue workplace settings and the effects of lisdexamfetamine dimesylate includes office-based tasks similar to school seat work. Unfortunately, this is inconsistent with the typical work environment most common for individuals with disabilities such as ADHD where food preparation is the most common job following high school. Therefore, medication effects in this type of setting, most common for individuals with ADHD entering the workforce, need to be studied. The investigators propose to study workplace behavior in an analogue work setting in a laboratory "pizza place." Individuals with ADHD will participate in an interview with a supervisor each day, have a list of deliveries that need to be managed, deal with situations that require occupational judgment and appropriate customer service, and drive to make deliveries accurately and on-time. These behaviors can be reliably assessed within the laboratory. Twenty young adults will participate in two "workdays" within a randomized, double-blind, placebo-controlled design wherein participants will be administered placebo and .3 mg/kg lisdexamfetamine dimesylate in a counter-balanced order.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ADHD
* parental permission and/or teen consent/assent as appropriate
* between 16-25 years of age
* IQ greater than or equal to 70
* permit or license to drive
* ability to read and understand English

Exclusion Criteria:

* any medical condition that would contraindicate use of stimulant medication
* any prior adverse response to lisdexamfetamine dimesylate or other stimulant medication
* use of concurrent,non-stimulant psychoactive medication
* diagnosis of schizophrenia or presence of thought disorder symptoms
* autism spectrum disorder

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordon CT, Fabiano GA, Hulme KF, Sodano SM, Adragna M, Lim R, Stanford S, Janikowski L, Bufalo B, Rodriguez Z, Swiatek D. Efficacy of lisdexamfetamine dimesylate for promoting occupational success in adolescents and young adults with attention-deficit/hyperactivity disorder. Exp Clin Psychopharmacol. 2021 Aug;29(4):308-318. doi: 10.1037/pha0000365. Epub 2020 Apr 16. PMID 32297783

RESULTS

PARTICIPANT FLOW:
Groups:
- Allocated to Vyvanse First: Administration of Vyvanse 40 mg then placebo on different days in a cross-over design
- Allocated to Placebo First: Allocated to placebo then Vyvanse 40 mg on different days
Period: Overall Study
Arm/Group | Allocated to Vyvanse First | Allocated to Placebo First
Started | 12 | 10
Completed | 10 | 10
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Did not complete entire visit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ADHD Participant: Administration of placebo capsule/Vyvanse 40 mg on different days in a cross-over design
Arm/Group | ADHD Participant
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.76 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Currently prescribed stimulant medication [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Ratings of Job Application Quality
Description: Three independent coders will review each de-identified application. Following the review of the application, coders will complete a rating form that asks them to make an overall evaluation regarding whether the person was an acceptable job candidate for an interview using a scale of 1 ("definitely not") to 5 ("definitely"). Average rating across coders will be used as the dependent measure.
Time Frame: during interventional study session, 1 day in duration
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Placebo
- Vyvanse: 40 mg Vyvanse
Arm/Group | Placebo | Vyvanse
Number analyzed (Participants) | 20 | 20
score on a scale | 3.40 (1.03) | 3.56 (1.00)

2. Primary Outcome: Ratings of Job Interview Performance
Description: Three coders who are unaware of the study participant identities or group status will view the job interview videotape and completed a form. Raters will provide a rating of their overall impression of the interview behavior ranging from a score of one (Poor) to four (Outstanding). The average score of the coders will be utilized as a dependent measure.
Time Frame: during interventional study session, 1 day in duration
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo; Vyvanse: 40 mg of Vyvanse administered q.a.m. or Placebo administered in random, counter-balanced fashion.
  Lisdexamfetamine Dimesylate 40 MG: Lisdexamfetamine Dimesylate 40 MG administered orally
  Placebo: Placebo capsule administered orally
Arm/Group | Placebo | Vyvanse
Number analyzed (Participants) | 20 | 20
score on a scale | 3.17 (.76) | 3.33 (.91)

3. Primary Outcome: Objective Observation of Workplace Productivity
Description: The dependent measures from this aspect of the study are the number of items completed correctly out of the total number of assigned items (i.e., 225). Thus, the score reflects the percentage of items correctly completed out of the 225 assigned and scores could range from 0-100.
Time Frame: during interventional study session, 1 day in duration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vyvanse
Number analyzed (Participants) | 20 | 20
score on a scale | 65.60 (17.55) | 68.45 (15.60)

4. Primary Outcome: Inattentive/Overactive Rating
Description: In addition to ratings of the interview performance, the rater also will complete the five-item inattentive/overactive (I/O) factor of the Iowa Conners rating scale (Atkins, Pelham, & Licht, 1989; Loney & Milich, 1982; Pelham, Milich, Murphy, & Murphy, 1989). The five items are rated on a scale of Not at all (0) to Very Much (3) and the sum of these items represents the score. The dependent measure will be the score averaged across raters. Scores can range from 0-3 on each item, and the average score of the 5 items was used. Higher scores reflect greater inattentive/overactivity-related behaviors.
Time Frame: during interventional study session, 1 day in duration
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Vyvanse
Number analyzed (Participants) | 20 | 20
score on a scale | 2.13 (1.33) | 2.01 (1.28)

ADVERSE EVENTS:
Time Frame: Each condition in the study (i.e., placebo, Vyvanse) was administered on a single day, approximately one week apart, for each participant. Adverse events were evaluated for the day of administration of each condition.
Description: The definition was not different from clinicaltrials.gov definitions.
Arm/Group | Placebo | Vyvanse
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03446885/Prot_SAP_000.pdf